CLINICAL TRIAL: NCT02663050
Title: The Effect of Kinesio Taping Application for Dysmenorrhea: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Kinesio Taping Application for Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Mustafa Ozturk, M.D.,Obstetrics and Gynecology, Specialist, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mustafa
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Dysmenorrhea
Keywords: Dysmenorrhea; kinesio tape
MeSH Terms: conditions — Dysmenorrhea | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Kinesio taping group (Experimental): only Kinesio taping treatment group
  Interventions: Other: Kinesio taping
- NSAID treatment group (Active Comparator): only NSAIDs taking group
  Interventions: Drug: NSAID's
- Combination treatment group (Active Comparator): NSAIDs plus Kinesio taping group
  Interventions: Other: Kinesio taping; Drug: NSAID's

INTERVENTIONS:
Other: Kinesio taping — Patients will be taped for four days , ıt will start at the begining of the Dysmenorrhea
  Arms: Combination treatment group; Kinesio taping group
Drug: NSAID's — twice a daily
  Other Names: Diclophenac Potassium
  Arms: Combination treatment group; NSAID treatment group

SUMMARY:
Dysmenorrhea is a common symptom in daily practice of gynecology. Different kind of treatment strategies are being held. But invasive and pharmacological therapies have good outcome with systemic side effects. Kinesio taping is being widely used in different pain conditions. Kinesio taping is a noninvasive and nonpharmacological, easy-to-use intervention method which can be used in outpatient practice without systemic side effects.

DETAILED DESCRIPTION:
Dysmenorrhea is a kind of visceral pain that result of peritoneal irritation. It is so common in gynecological outpatient practice. Most of treatment is based pharmacological treatments as NSAIDs, oral contraceptives with many side effects. Kinesio taping is widely used for musculoskeletal parenchymal pain like sports related injuries. As in other complementary treatment methods like acupuncture and acupressure; pain carrying unmyelinated thin pain fibers are blocked by touch sensation carrying myelinated thick fibers which is stimulated by acupressure(gate control theory by Melzack), kinesio taping blocks the pain fibers that comes from same spinal level. So it can be used easily and instantly for dismenore

ELIGIBILITY:
Inclusion Criteria:

* Dysmenorrhea

Exclusion Criteria:

* pregnancy
* surgical abdominal emergency
* metabolic or inflammatory illnesses or cardiovascular diseases,
* endocrine disorders such as diabetes, thyroid disorders, androgen excess (hyperprolactinemia, uncontrolled thyroid disease, congenital adrenal hyperplasia, Cushing's syndrome, androgen-secreting tumor),
* smokers
* using pharmaceutical agents such as anti-inflammatory agents that could possibly impact on endocrine and liver enzymes
* musculoskeletal pain
* inguinal hernia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | 0- 4th day
  At the begining of the Dysmenorrhea before taping we will measure the VAS level (pretreatment)and 4 days after taping we will measure the second VAS level (after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Öztürk, M.D., Principal Investigator — Etimesgut Military Hospital

IPD SHARING:
Plan to Share IPD: Yes
We will share the data monthly